CLINICAL TRIAL: NCT05428423
Title: Assessment of the Reliability of Changes in Plethysmography Variability Index During Tidal Volume Challenge for Predicting Fluid Responsiveness in Intensive Care Unit Patients
Brief Title: Reliability of PVI Changes During Tidal Volume Challenge in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Xavier Monnet, Professor, Bicetre Hospital
Other Study IDs: IDRCB:2022-A01253-40
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Shock; Septic Shock; Sepsis; Hemodynamic Instability
Keywords: Tidal volume challenge; Pleth variability index
MeSH Terms: conditions — Shock; Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess whether changes in the plethysmography variability index, during a tidal volume challenge, can reliably detect simultaneous changes in arterial blood pressure pulsatility, in patients hospitalized in intensive care unit. If results will be positive, this will allow the test to be performed even in the absence of an invasive arterial catheter.

DETAILED DESCRIPTION:
Among patients in a state of shock one of the first treatments is volume expansion, consisting in a fast intravenous injection of crystalloid or colloid solutions in order to increase cardiac preload and consequently cardiac output. However, this augmentation of the cardiac output happens only in half of the patients.To avoid ineffective fluid administration several tests have been developed.

One of these tests is called the "tidal volume challenge" (TVC). It consists of transiently increasing for 1 minute the volume of air inhaled with each breath, in mechanically ventilated patients, and then evaluating whether this change impacts the pulsatility of the arterial blood pressure, detected by an arterial catheter. This test seems reliable, but it requires an arterial catheter to be in place.

It has been suggested in previous studies that pulsatility of blood pressure can be estimated by the pulsatility of the plethysmography signal ("plethysmography variability index"), obtained from the oxygen saturation signal that's measured in all intensive care patients. The advantage is that this measurement only requires a sensor placed at the end of a finger, on the earlobe or on the forehead.

The aim of the study is to assess whether changes in the plethysmography variability index (PVI) during a TVC can reliably detect simultaneous changes in blood pressure pulsatility. This study will include patients hospitalized in intensive care unit, mechanically ventilated, in whom physicians have decided to perform a TVC as common practice. Changes, occurred during this test, in arterial blood pressure pulsatility and in plethysmography pulsatility index will be measured and compared. If results will show that changes in PVI during TVC are reliable for measuring blood pressure pulsatility changes during this test, this will allow the test to be used even in the absence of an arterial catheter.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in intensive care unit
* physicians' decision to perform a tidal volume challenge
* hemodynamic monitoring with a calibrated pulse contour analysis device (PICCO2) in place
* monitoring of oxygen saturation with Masimo SET
* mechanical ventilation with tidal volume of 6 ml/kg on ideal body weight

Exclusion Criteria:

* thoracic drainage
* patient under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized in intensive care unit, mechanically ventilated with a tidal volume of 6 ml/kg on ideal body weight, with oxygen saturation monitoring with Masimo SET and cardiac output monitoring with PICCO2 system in place.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Reliability of PVI changes in diagnosing preload responsiveness during TVC | TVC is performed in 1 minute
  The primary objective is to assess the reliability of PVI changes induced by a tidal volume challenge test in diagnosing a preload responsiveness state in adult ICU patients.

SECONDARY OUTCOMES:
Reliability of PVI absolute values to diagnose preload responsiveness | TVC is performed in 1 minute
  Secondary objective is to test the reliability of absolute values of PVI to diagnose a preload responsiveness state in adult intensive care patients.
Evaluation of PVI changes during TVC according to sensor position | TVC is performed in 1 minute
  Third objective is to compare the value of changes in PVI induced by a tidal volume challenge test to diagnose a preload responsiveness state according to the location of the plethysmographic measurement (finger, earlobe, forehead).
Comparison of PPV and PVI changes during PLR test or volume expansion | PLR is performed in 1 minute
  Forth objective is to compare the changes in pulse pressure variation (PPV) and PVI during a passive leg raising test (PLR) and a volume expansion, if applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Monnet, MD-PhD, Principal Investigator — Hopital de Bicetre
Locations (1):
- Service de médecine intensive-réanimation, Hôpital de Bicêtre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Background] Marik PE, Monnet X, Teboul JL. Hemodynamic parameters to guide fluid therapy. Ann Intensive Care. 2011 Mar 21;1(1):1. doi: 10.1186/2110-5820-1-1. PMID 21906322
- [Background] National Heart, Lung, and Blood Institute Acute Respiratory Distress Syndrome (ARDS) Clinical Trials Network; Wiedemann HP, Wheeler AP, Bernard GR, Thompson BT, Hayden D, deBoisblanc B, Connors AF Jr, Hite RD, Harabin AL. Comparison of two fluid-management strategies in acute lung injury. N Engl J Med. 2006 Jun 15;354(24):2564-75. doi: 10.1056/NEJMoa062200. Epub 2006 May 21. PMID 16714767
- [Background] Myatra SN, Prabu NR, Divatia JV, Monnet X, Kulkarni AP, Teboul JL. The Changes in Pulse Pressure Variation or Stroke Volume Variation After a "Tidal Volume Challenge" Reliably Predict Fluid Responsiveness During Low Tidal Volume Ventilation. Crit Care Med. 2017 Mar;45(3):415-421. doi: 10.1097/CCM.0000000000002183. PMID 27922879
- [Background] Alvarado Sanchez JI, Caicedo Ruiz JD, Diaztagle Fernandez JJ, Amaya Zuniga WF, Ospina-Tascon GA, Cruz Martinez LE. Predictors of fluid responsiveness in critically ill patients mechanically ventilated at low tidal volumes: systematic review and meta-analysis. Ann Intensive Care. 2021 Feb 8;11(1):28. doi: 10.1186/s13613-021-00817-5. PMID 33555488
- [Background] Feissel M, Teboul JL, Merlani P, Badie J, Faller JP, Bendjelid K. Plethysmographic dynamic indices predict fluid responsiveness in septic ventilated patients. Intensive Care Med. 2007 Jun;33(6):993-9. doi: 10.1007/s00134-007-0602-6. Epub 2007 Mar 29. PMID 17393139
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Natalini G, Rosano A, Taranto M, Faggian B, Vittorielli E, Bernardini A. Arterial versus plethysmographic dynamic indices to test responsiveness for testing fluid administration in hypotensive patients: a clinical trial. Anesth Analg. 2006 Dec;103(6):1478-84. doi: 10.1213/01.ane.0000246811.88524.75. PMID 17122227
- [Background] Cannesson M, Attof Y, Rosamel P, Desebbe O, Joseph P, Metton O, Bastien O, Lehot JJ. Respiratory variations in pulse oximetry plethysmographic waveform amplitude to predict fluid responsiveness in the operating room. Anesthesiology. 2007 Jun;106(6):1105-11. doi: 10.1097/01.anes.0000267593.72744.20. PMID 17525584
- [Background] Cannesson M, Desebbe O, Hachemi M, Jacques D, Bastien O, Lehot JJ. Respiratory variations in pulse oximeter waveform amplitude are influenced by venous return in mechanically ventilated patients under general anaesthesia. Eur J Anaesthesiol. 2007 Mar;24(3):245-51. doi: 10.1017/S026502150600161X. Epub 2006 Oct 23. PMID 17054816
- [Background] Cannesson M, Desebbe O, Rosamel P, Delannoy B, Robin J, Bastien O, Lehot JJ. Pleth variability index to monitor the respiratory variations in the pulse oximeter plethysmographic waveform amplitude and predict fluid responsiveness in the operating theatre. Br J Anaesth. 2008 Aug;101(2):200-6. doi: 10.1093/bja/aen133. Epub 2008 Jun 2. PMID 18522935
- [Background] Landsverk SA, Hoiseth LO, Kvandal P, Hisdal J, Skare O, Kirkeboen KA. Poor agreement between respiratory variations in pulse oximetry photoplethysmographic waveform amplitude and pulse pressure in intensive care unit patients. Anesthesiology. 2008 Nov;109(5):849-55. doi: 10.1097/ALN.0b013e3181895f9f. PMID 18946297
- [Background] Liu T, Xu C, Wang M, Niu Z, Qi D. Reliability of pleth variability index in predicting preload responsiveness of mechanically ventilated patients under various conditions: a systematic review and meta-analysis. BMC Anesthesiol. 2019 May 8;19(1):67. doi: 10.1186/s12871-019-0744-4. PMID 31068139
- [Background] Monnet X, Guerin L, Jozwiak M, Bataille A, Julien F, Richard C, Teboul JL. Pleth variability index is a weak predictor of fluid responsiveness in patients receiving norepinephrine. Br J Anaesth. 2013 Feb;110(2):207-13. doi: 10.1093/bja/aes373. Epub 2012 Oct 26. PMID 23103777
- [Background] Coeckelenbergh S, Delaporte A, Ghoundiwal D, Bidgoli J, Fils JF, Schmartz D, Van der Linden P. Pleth variability index versus pulse pressure variation for intraoperative goal-directed fluid therapy in patients undergoing low-to-moderate risk abdominal surgery: a randomized controlled trial. BMC Anesthesiol. 2019 Mar 9;19(1):34. doi: 10.1186/s12871-019-0707-9. PMID 30851740
- [Background] Taccheri T, Gavelli F, Teboul JL, Shi R, Monnet X. Do changes in pulse pressure variation and inferior vena cava distensibility during passive leg raising and tidal volume challenge detect preload responsiveness in case of low tidal volume ventilation? Crit Care. 2021 Mar 18;25(1):110. doi: 10.1186/s13054-021-03515-7. PMID 33736672